CLINICAL TRIAL: NCT06141746
Title: Ultrasound Assessment of Irrigation Fluid Effect on Extravascular Lung Water in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Ultrasound Assessment of Extravascular Lung Water in Patients Undergoing Percutaneous Nephrolithotomy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Ahmed Hashem, Principal investigator, Assiut University
Other Study IDs: Extravascular lung water
Record Dates: First submitted 2023-10-20; First posted 2023-11-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Extravascular Lung Water; Percutaneous Nephrolithotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lung ultrasound — Early detection of fluid accumulation in alveolar, interstitial and intracellular compartments of the lung due to intravascular absorption of irrigation fluid of PNL guided by lung ultrasound by detection of sonographic B lines.

SUMMARY:
Early detection of fluid accumulation in alveolar, interstitial and intracellular compartments of the lung due to intravascular absorption of irrigation fluid of PNL guided by lung ultrasound by detection of sonographic B lines.

DETAILED DESCRIPTION:
Study protocol:

Anesthetic technique:- After adequate pre-oxygenation for 3-5 min, General anesthesia will be induced by intravenous lidocaine 60 mg, propofol (2mg/kg) and cis-atracurium (0.15 mg/ kg) to facilitate endotracheal intubation by a cuffed endotracheal tube (size 6.5-7.5-mm), then the patient will be connected to mechanical ventilation which will be maintained with an 8 ml/ kg tidal volume, and ventilation frequency well be adjusted to maintain end-tidal CO2 between 30-35 mmHg. Anesthesia will be maintained with isoflurane (0.8-1.0%) in a mixture of oxygen and air (50:50%) and cis-atracurium (0.03 mg/ kg) and maintained every 20 min. Standard monitoring will be used intraoperatively including non-invasive arterial blood pressure, electrocardiography, end-tidal CO2, peripheral oxygen saturation and esophageal core temperature. Patients will receive one liter of normal saline infused over the first 2 hours intraoperatively as their fasting requirements and will be infused with 3 ml/kg/hour of Ringer's acetate as a maintenance fluid. Intraoperative hypotension (more than 20% decrease of the baseline of the patient ) will be treated by a bolus dose of crystalloid (4 ml/kg) as well as a bolus dose of ephedrine (3 mg). Atropine (0.5 mg) will be used to treat bradycardia if the heart rate is <60 beat/min. At end of surgery, isoflurane will be discontinued, and neuromuscular block will be antagonized using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), intravenous paracetamol will be given as analgesia and boluses of fentanil Intraoperative as needed . Extubation will performed when patients began breathing spontaneously and were able to respond to verbal requests and discharge to post-Anesthesia Care Unit (PACU) but if the patient is not fulfilling criteria of extubation so discharge will be to Intensive care unit (ICU). If acute Postoperative lung congestion occurs with postoperative hypoxemia and desaturation, it will be treated with furosemide.

Blood samples will be collected for CBC, ABG and electrolytes as sodium and potassium Pre-operative, intraoperative and Immediately Post-operative.

Lung ultrasound scan technique: -

Each patient will be assessed for the presence of B-lines before induction of anesthesia and after end of anesthesia. A curved 2-6-MHz probe of Mindray machine will be used to do a series of scans with the patient in the supine position by applying the probe perpendicular to the skin over intercostal spaces along anatomical reference lines. More precisely, we will scan the anterolateral hemithoraxes along the parasternal, midclavicular, anterior axillary and mid-axillary lines. The left hemithorax will be scanned from the second to the fourth intercostal space, whereas the right lung will be scanned from the second to the fifth intercostal space, giving a total of 28 scanning sites. The edematous lung shows B-lines as vertical narrow bands originating from the pleural line and extending to the bottom of the image. A B-line score of ≤5 will be considered a normal sonographic pattern, since a few B-lines can be present in healthy subjects, especially above the diaphragm.

Data collection:- Patient characteristics

* Age
* Sex
* Medical disease
* Drug intake Operative data
* Mean arterial blood pressure (MAP), heart rate and peripheral oxygen saturation during the following times (before induction of anesthesia, every 15 minutes after intubation, and at the end of surgery)
* Intraoperative complication and interventions.
* Duration of surgery
* Duration of anesthesia
* Type, volume and height of irrigation fluid.
* Ultrasound guided extravascular lung water.

Postoperative data

* Hemoglobin assessment.
* Serum sodium level.
* Serum potassium level.
* Arterial blood gases (ABG).
* Ultrasound guided extravascular lung water.

Statistical analysis:-

●Descriptive analysis Statistical analysis will be carried out by the SPSS statistical software package version 26.0 (IBM/SPSS, Inc., Chicago, IL). Baseline characteristics will be defined using descriptive statistics. Categorical variables were stated as an absolute number (n) and a relative frequency (%), and continuous variables will be represented as a median (interquartile range) or as a mean (± SD), depending on the normality of the distribution. The normality of distribution will be tested by the one-sample Kolmogorov-Smirnov test.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class I, II or III adult patients of age group 18-65 years. •Patient undergoing percutaneous nephrolithotomy.

Exclusion Criteria:

* •Patients unable to provide written consent.

  * Patients less than 18 years or above 65 years.
  * ASA Class IV.
  * Patients previously diagnosed to suffer from interstitial lung disease.
  * patients who will receive intraoperative diuretics

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be carried on patients who are undergoing percutaneous nephrolithotomy under general anesthesia between Nov.2023 and Nov.2024.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lung congestion | 1 hour postoperative
  Incidence of Post-operative lung congestion quantified by number of sonographic B-lines in anterolateral lung ultrasound scan in patients undergoing percutaneous nephrolithotomy.

SECONDARY OUTCOMES:
Immediately Post-operative and after 24hours postoperative hemoglobin assessment. | 1 hour postoperative
  Immediately Post-operative and after 24hours postoperative hemoglobin assessment.
Immediately Post-operative and after 24hours postoperative serum sodium and potassium assessment. | 1 hour postoperative
  Immediately Post-operative and after 24hours postoperative serum sodium and potassium assessment.
Immediately Post-operative and after 24hours postoperative arterial blood gases (ABG) assessment. | 1 hour postoperative
  Immediately Post-operative and after 24hours postoperative arterial blood gases (ABG) assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ezzat, Study Director — Assiut University

REFERENCES:
- [Background] Romero V, Akpinar H, Assimos DG. Kidney stones: a global picture of prevalence, incidence, and associated risk factors. Rev Urol. 2010 Spring;12(2-3):e86-96. PMID 20811557
- [Background] De S, Autorino R, Kim FJ, Zargar H, Laydner H, Balsamo R, Torricelli FC, Di Palma C, Molina WR, Monga M, De Sio M. Percutaneous nephrolithotomy versus retrograde intrarenal surgery: a systematic review and meta-analysis. Eur Urol. 2015 Jan;67(1):125-137. doi: 10.1016/j.eururo.2014.07.003. Epub 2014 Jul 23. PMID 25064687
- [Background] Rozentsveig V, Neulander EZ, Roussabrov E, Schwartz A, Lismer L, Gurevich B, Klein Y, Weksler N. Anesthetic considerations during percutaneous nephrolithotomy. J Clin Anesth. 2007 Aug;19(5):351-5. doi: 10.1016/j.jclinane.2007.02.010. PMID 17869985
- [Background] Gehring H, Nahm W, Zimmermann K, Fornara P, Ocklitz E, Schmucker P. Irrigating fluid absorption during percutaneous nephrolithotripsy. Acta Anaesthesiol Scand. 1999 Mar;43(3):316-21. doi: 10.1034/j.1399-6576.1999.430312.x. PMID 10081538
- [Background] Kukreja RA, Desai MR, Sabnis RB, Patel SH. Fluid absorption during percutaneous nephrolithotomy: does it matter? J Endourol. 2002 May;16(4):221-4. doi: 10.1089/089277902753752160. PMID 12042103
- [Background] Atici S, Zeren S, Aribogan A. Hormonal and hemodynamic changes during percutaneous nephrolithotomy. Int Urol Nephrol. 2001;32(3):311-4. doi: 10.1023/a:1017527126481. PMID 11583340
- [Background] Koroglu A, Togal T, Cicek M, Kilic S, Ayas A, Ersoy MO. The effects of irrigation fluid volume and irrigation time on fluid electrolyte balance and hemodynamics in percutaneous nephrolithotripsy. Int Urol Nephrol. 2003;35(1):1-6. doi: 10.1023/a:1025956810783. PMID 14620272
- [Background] Mohta M, Bhagchandani T, Tyagi A, Pendse M, Sethi AK. Haemodynamic, electrolyte and metabolic changes during percutaneous nephrolithotomy. Int Urol Nephrol. 2008;40(2):477-82. doi: 10.1007/s11255-006-9093-6. PMID 17318347
- [Background] Cordts PR, LaMorte WW, Fisher JB, DelGuercio C, Niehoff J, Pivacek LE, Dennis RC, Siebens H, Georgio A, Valeri CR, et al. Poor predictive value of hematocrit and hemodynamic parameters for erythrocyte deficits after extensive elective vascular operations. Surg Gynecol Obstet. 1992 Sep;175(3):243-8. PMID 1514159
- [Background] Grathwohl KW, Bruns BJ, LeBrun CJ, Ohno AK, Dillard TA, Cushner HM. Does hemodilution exist? Effects of saline infusion on hematologic parameters in euvolemic subjects. South Med J. 1996 Jan;89(1):51-5. doi: 10.1097/00007611-199601000-00008. PMID 8545692
- [Background] Guzelburc V, Balasar M, Colakogullari M, Guven S, Kandemir A, Ozturk A, Karaaslan P, Erkurt B, Albayrak S. Comparison of absorbed irrigation fluid volumes during retrograde intrarenal surgery and percutaneous nephrolithotomy for the treatment of kidney stones larger than 2 cm. Springerplus. 2016 Oct 4;5(1):1707. doi: 10.1186/s40064-016-3383-y. eCollection 2016. PMID 27757377
- [Background] Wang CH, Chen NC, Tsai MS, Yu PH, Wang AY, Chang WT, Huang CH, Chen WJ. Therapeutic Hypothermia and the Risk of Hemorrhage: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Medicine (Baltimore). 2015 Nov;94(47):e2152. doi: 10.1097/MD.0000000000002152. PMID 26632746
- [Background] Shin HJ, Na HS, Jeon YT, Park HP, Nam SW, Hwang JW. The impact of irrigating fluid absorption on blood coagulation in patients undergoing transurethral resection of the prostate: A prospective observational study using rotational thromboelastometry. Medicine (Baltimore). 2017 Jan;96(2):e5468. doi: 10.1097/MD.0000000000005468. PMID 28079789